CLINICAL TRIAL: NCT06517017
Title: Use of Isatuximab, Dexamethasone and Lenalidomide in a Go-Slow Fashion for Ultra-Frail Patients With Multiple Myeloma: A Phase 2 Multicenter Study
Brief Title: Use of Isatuximab, Dexamethasone and Lenalidomide in a Go-Slow Fashion for Ultra-Frail Patients With Multiple Myeloma
Acronym: UltraFrailMM
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Utah (Other)
Collaborators: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HCI171326
Record Dates: First submitted 2024-07-12; First posted 2024-07-24 (Actual); Last update posted 2025-11-28 (Actual); Status verified 2025-11

CONDITIONS: Multiple Myeloma; Plasma Cell Leukemia
MeSH Terms: conditions — Multiple Myeloma; Leukemia, Plasma Cell | interventions — isatuximab; Dexamethasone; Lenalidomide

STUDY DESIGN:
Intervention Model Description: This is a single arm phase 2 study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Combination Treatment (Experimental): Isatuximab
  Interventions: Drug: Isatuximab

INTERVENTIONS:
Drug: Isatuximab — Subcutaneous isatuximab will be administered weekly on a 28-day cycle during the first two cycles, and every two weeks of a 28-day cycle thereafter. Dexamethasone will be administered on the days of isatuximab administration and can be discontinued after two cycles of therapy, or continued at discretion of investigator. Lenalidomide, will be added after two cycles of therapy have been completed.
  Other Names: Dexamethasone; Lenalidomide

SUMMARY:
Historically, the frailest patients with multiple myeloma are under-represented in clinical trials, and have very high rates of treatment discontinuation, and early treatment mortality. The investigators hypothesize that a go-slow gentle approach to starting treatment in such patients, starting with just Isatuximab and dexamethasone with a gentle introduction to lenalidomide third cycle onwards, may improve treatment adherence and quality of life. The goal of this clinical trial is to learn if a go-slow approach to treating MM in ultra-frail patients may improve the ability to adhere to treatment and improve quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subject aged ≥ 18 years.
* Histologically confirmed myeloma and/or Plasma Cell Leukemia who are newly diagnosed and having completed ≤ 1 prior cycle of myeloma treatment.
* For female subjects of childbearing potential: Negative pregnancy test or evidence of post-menopausal status or evidence of permanent surgical sterilization (bilateral oophorectomy or hysterectomy). The post-menopausal status will be defined as having been amenorrheic for 24 months without an alternative medical cause.
* Subjects must be willing to follow contraception requirements listed in the protocol, agree to participate in the Lenalidomide REMS program, and have signed the Patient-Physician Agreement Form.
* Male subjects must agree to use a latex condom during intercourse for the duration of study therapy as described in the protocol, even if he has undergone a successful vasectomy.
* Recovery to baseline or ≤ Grade 1 CTCAE v5 from toxicities related to any prior treatments, unless AE(s) are clinically nonsignificant and/or stable on supportive therapy per the treating investigator.
* Able to provide informed consent and willing to sign an approved consent form that conforms to federal and institutional guidelines.
* IMWG defined frailty score ≥ 3. IMWG definition available here: http://www.myelomafrailtyscorecalculator.net

Exclusion Criteria:

* Receiving other investigational agents.
* Any condition that would, in the Investigator's judgment, compromise the subject's ability to understand the subject information, give informed consent, and/or contraindicate the subject's participation in the clinical study due to safety concerns or compliance with clinical study procedures (e.g., infection/inflammation, intestinal obstruction, unable to swallow medication, [subjects may not receive the drug through a feeding tube], social/ psychological issues, etc.)
* Known prior severe hypersensitivity (NCI CTCAE v5.0 Grade ≥ 3) to investigational product (IP) or any component in its formulations. This includes hypersensitivity or history of intolerance to steroids, mannitol, pregelatinized starch, sodium stearyl fumarate, histidine (as base and hydrochloride salt), arginine hydrochloride, poloxamer 188, sucrose or any of the other components of study intervention that are not amenable to premedication with steroids and H2 blockers or would prohibit further treatment with these agents.
* Subjects currently taking prohibited medications as described in the protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-10-09 (Actual); Primary Completion 2026-11 (Estimated); Study Completion 2027-11 (Estimated)

PRIMARY OUTCOMES:
Completion rate of 9 cycles of treatment | At the end of 9 cycles of treatment (each cycle is 28 days)
  Assess the feasibility of approach incorporating the use of isatuximab and dexamethasone with the subsequent addition of lenalidomide from the third cycle onwards in ultra-frail patients with myeloma

SECONDARY OUTCOMES:
Change in quality of life as per the European Organization for Research and Treatment of Cancer Quality of Life Questionnaire C30 domain | At the end of 4 cycles of treatment (each cycle is 28 days)
  Assess if an approach incorporating the use of isatuximab and dexamethasone with the subsequent addition of a lenalidomide in ultra-frail patients with myeloma leads to an improvement in quality of life as measured by the EORTC score. The questionnaire has 10 subscales, each with a score range of 0 to 100 points. Higher scores on the functional scales and global quality of life indicate better functioning, while higher scores on the symptom scales indicate a higher symptom burden. The QLQ-C30 summary score is calculated by averaging the scores of the 13 scales and items, with a higher score indicating a better health-related quality of life (HRQoL).
Frequency of adverse events (AEs) and serious adverse events (SAEs) characterized by type | At study completion. Participants will be enrolled in study for about 3 years.
  Assess the safety and tolerability of isatuximab, lenalidomide and dexamethasone in the study population.
Frequency of adverse events (AEs) and serious adverse events (SAEs) characterized by severity (as defined by the NIH CTCAE, version 5.0) | At study completion. Participants will be enrolled in study for about 3 years.
  Assess the safety and tolerability of isatuximab, lenalidomide and dexamethasone in the study population.
Frequency of adverse events (AEs) and serious adverse events (SAEs) characterized by seriousness | At study completion. Participants will be enrolled in study for about 3 years.
  Assess the safety and tolerability of isatuximab, lenalidomide and dexamethasone in the study population.
Frequency of adverse events (AEs) and serious adverse events (SAEs) characterized by duration | At study completion. Participants will be enrolled in study for about 3 years.
  Assess the safety and tolerability of isatuximab, lenalidomide and dexamethasone in the study population.
Frequency of adverse events (AEs) and serious adverse events (SAEs) characterized by relationship to study treatment | At study completion. Participants will be enrolled in study for about 3 years.
  Assess the safety and tolerability of isatuximab, lenalidomide and dexamethasone in the study population.
Overall survival (OS) | Time from registration until 3 years from start of therapy or death from any cause.
  Assess overall survival in this study population

CONTACTS AND LOCATIONS:
Overall Officials: Ghulam Rehman Mohyuddin, MBBS, Principal Investigator — Huntsman Cancer Institute
Locations (1):
- Huntsman Cancer Institute at the University of Utah, Salt Lake City, Utah, United States

IPD SHARING:
Plan to Share IPD: No